CLINICAL TRIAL: NCT04322071
Title: Factors Affecting Diabetes Self-management in Young People and Their Families: a Qualitative Study
Brief Title: Family Factors in Young People With Diabetes: a Qualitative Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Southampton (Other)
Collaborators: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 52030
Record Dates: First submitted 2020-03-04; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Type 1 Diabetes
Keywords: Children and young people; Family; Qualitative
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lower risk of long term complications: Young people with diabetes who have HbA1c <58mmols/mol, and family members.
  Interventions: Other: Interview
- Higher risk of long term complications: Young people with diabetes who have HbA1c ≥75mmols/mol and <100mmols/mol, and family members.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Qualitative interviews only

SUMMARY:
8 young people (aged 12-15yrs) with type 1 diabetes will be interviewed along with their families during this qualitative study. The interviews will explore factors identified by the young people and their families as important in diabetes management. Comparison of these factors will then be made between the young people with higher and lower HbA1c levels.

DETAILED DESCRIPTION:
Family is an important factor in the self-management of type 1 diabetes by children and young people. Existing research has explored the experience of living with diabetes, considered from the perspective of children and parents, but has not provided children's diabetes teams with the information they need to support young people with higher blood glucose levels, and therefore higher risks of long term complications related to their diabetes.

During this qualitative study the researcher will meet with young people (aged 12-15yrs) and their families for a joint interview, held in the family home, exploring the factors which they consider important in diabetes self-management.

One interview will be held with each family. Recruitment of 8 families is planned.

The interviews will be recorded and transcribed to allow thematic analysis, allowing identification of common factors considered to be important by families.

The HbA1c of young people with diabetes is checked regularly in clinic and provides an assessment of blood glucose levels over the preceding months. Higher HbA1c levels are associated with higher risk of long term complications.

The index young people will be recruited in 2 groups: one group will have lower risk of long term complications (identified by an HbA1c level of <58mmol/mol). The other will have higher risk (HbA1c 75-100mmol/mol). A comparison will be made between the families in each group, to identify which themes are more common in the lower or higher risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 - 15 years (between their 12th and 16th birthday at recruitment)
* Type 1 diabetes diagnosed for at least 6 months
* Group 1: HbA1c <58mmols/mol on last known test
* Group 2: HbA1c ≥75mmols/mol and <100mmols/mol on last known test
* Willing to participate in group interview with at least one parent/carer

Exclusion Criteria:

* Family currently identified as not suitable for lone visits
* Participants with inadequate English to take part in a semi-structured interview conducted in English
* Children and Young people for whom the last HbA1c incongruent with their previous results will be excluded

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Young people aged 12-15yrs with HbA1c in one of the two groups (4 from each group) will be identified from the caseload of the East Kent Children's Diabetes Team. They will be invited to participate in interviews along with at least one parent/carer, and up to 4 other people (including children) which they identify as important in their diabetes management.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Thematic Analysis | Interviews of up to 90mins conducted during the study period (a period of 5 weeks ending on the 31st of March 2020)
  Themes identified against the primary question: what factors do families identify as important in self-management of a young person's Type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Anitha Kumaran, MBBS, PhD, Principal Investigator — University of Southampton
Locations (1):
- East Kent Hospitals University Foundation NHS Trust, Ashford, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No